CLINICAL TRIAL: NCT03580382
Title: Study of CDX-3379, a Human Monoclonal Antibody Targeting ERBB3, in Combination With the MEK Inhibitor, Trametinib, in Patients With Advanced Stage NRAS Mutant and BRAF/NRAS Wildtype (WT) Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per regulatory coordinator, the sponsor is no longer supporting the study.
Sponsor: NYU Langone Health (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00363
Record Dates: First submitted 2018-07-05; First posted 2018-07-09 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRAS mutant melanoma (Experimental): C1D1-C1D21, CDX-3379 D1Trametinib daily Biopsy (days 14-16)
  Interventions: Drug: Trametinib daily Until PD; Drug: CDX-3379 (ERBB3 antibody)
- WT melanoma (Experimental): C1D1-C1D21, CDX-3379 D1Trametinib daily Biopsy (days 14-16)
  Interventions: Drug: Trametinib daily Until PD; Drug: CDX-3379 (ERBB3 antibody)

INTERVENTIONS:
Drug: Trametinib daily Until PD — 1.0 mg daily
Drug: CDX-3379 (ERBB3 antibody) — 15mg/kg IV Q3W

SUMMARY:
The main goal of this study is to test if it is safe and effective to give CDX-3379 together to treat advanced melanoma in patients with the NRAS mutation and BRAF/NRAS wildtype.

DETAILED DESCRIPTION:
Primary Objectives:

Phase 1b: To determine the RP2D and assess the toxicity and tolerability of the combination of CDX-3379 (ERBB3 antibody) and trametinib (MEK inhibitor) in NRAS and BRAF/NRAS WT melanoma patients

Phase 2: To estimate the response rates and duration of response of the combination of CDX-3379 (ERBB3 antibody) and trametinib in NRAS positive and BRAF/NRAS WT melanoma patients

Secondary/Exploratory Objectives:

Phase 1b: To assess clinical activity and steady-state pharmacokinetics of CDX-3379 and trametinib Phase 2: To compare the efficacy of the combination of CDX-3379 (ERBB3 antibody) and trametinib is more effective than a MEK inhibitor alone in NRAS positive and BRAF/NRAS WT melanoma patients alone using locally assessed progression free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Read, understood, and provided written informed consent and, if applicable, Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures.

  2. Male or female patients who are 18 years of age or older. 3. Patients with a diagnosis of histologically confirmed advanced (defined as unresectable stage III or IV) melanoma with the NRAS Q61 mutation or BRAF/NRAS WT for which there is no remaining standard therapy with curative potential or patients are ineligible or unable to tolerate therapy with curative potential.
  * Any standard of care mutation testing is acceptable to document mutation status.

    4.Patients must have archival tissue and at least one disease site amenable to biopsy:
  * For phase Ib, all patients will undergo fresh tumor biopsy
  * For phase II, five patients with NRAS mutation and five patients with BRAF/NRAS WT melanoma will undergo fresh tumor biopsy 5.Measurable (target) disease by Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Target lesions selected for tumor measurements should be those where additional (eg palliative) treatments are not indicated or anticipated.
  * Measurable disease per RECIST 1.1 requirements: defined as longest diameter to be recorded for non-nodal lesions > 10mm and short axis for nodal lesions >15 mm using conventional techniques 6.All residual toxicity related to prior radiotherapy or anticancer therapies (excluding alopecia, grade 2 fatigue, vitiligo or endocrinopathies on stable replacement therapy) must resolve to grade 1 severity or less (or returned to baseline) prior to receipt of study treatment.

    7.Adequate electrolytes, liver, renal, and hematology function as defined below:

    a.Hemoglobin ≥ 9 g/dL b.Absolute neutrophil count ≥ 1500/mm3 c.Platelet count ≥ 100,000/mm3 d.Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) (≤ 5 × ULN for cases involving liver metastasis) e.Bilirubin ≤ 1.5 × ULN (≤ 5 × ULN for cases of documented or suspected Gilbert's disease) f.Serum creatinine ≤ 1.5 g/dL or calculated creatinine clearance (CrCl) ≥60 mL/min for patients with serum creatinine > 1.5 x ULN g.Serum magnesium, calcium and potassium within normal limits 8.Life expectancy ≥ 12 weeks 9.ECOG performance status (PS) < 1 10.Willing and able to comply with scheduled visits, treatment plan, and laboratory tests.

    11.Screening EKG without clinically significant abnormalities. 12.Corrected (Fridericia's) QTcF must be < 480 milliseconds. 13.Allowance of prior therapy regimens:
  * No limit on prior number of regimens
  * Must have completed prior cytotoxic chemotherapy a minimum of 4 weeks prior to starting study treatment (except for bis-chlorethynitrosurea (BCNU)), which must have been completed a minimum of 6 weeks prior to starting therapy.
  * Prior localized radiation therapy must have been completed a minimum of 2 weeks prior to starting therapy and the patient must have baseline imaging with a full body PET-CT or CT scans of the chest, abdomen, and pelvis and within 4 weeks prior to study enrollment.
  * For CNS metastases, disease must be treated and demonstrate stability with Brain MRI a minimum of 2 weeks prior to starting therapy.

    14.Both male and female patients enrolled in this trial must agree to use highly effective contraception during the course of the trial and for at least for 6 months after the final dose of CDX-3379 (an effective form of contraception is an oral contraceptive or a double barrier method), or greater, as in accordance with the label requirements for trametinib. Patients and/or partners who are surgically sterile or postmenopausal are exempt from this requirement.
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after stopping study drug. Highly effective contraception methods include:
  * Total abstinence or
  * Male or female sterilization or
  * Combination of any two of the following (a+b or a+c or b+c):

    1. Use of oral, injected or implanted hormonal methods of contraception; hormonal contraceptives are not acceptable as a sole method of contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository 15. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Exclusion Criteria:

1. Received CDX-3379 or other anti-ErbB3 targeted agents previously.
2. Received trametinib or other MEK inhibitor agents previously.
3. Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
4. Other prior malignancy active within 2 years, except for localized prostate cancer, cervical carcinoma in situ, non-melanomatous carcinoma of the skin, stage 1 differentiated thyroid cancer or ductal carcinoma in situ of the breast that has/have undergone curative surgery or radiation.
5. Active central nervous system (CNS) metastases are excluded. Known brain metastases must have been previously treated and asymptomatic for 2 weeks and not progressive in size or number for 4 weeks prior to enrollment, documented via scans. Continued use of anticonvulsants (in the absence of any suspicion of progressive brain metastases) is acceptable. Patients must currently be on a stable, lowest possible dose of steroids.
6. Radiation therapy within 14 days prior to the first scheduled dose in this study, including, in addition (if necessary), the timeframe for resolution of any actual or anticipated toxicities from such radiation.
7. Known HIV, hepatitis B or hepatitis C infection, or active infection requiring systemic intravenous therapy
8. Use of any monoclonal based therapies within 4 weeks (excluding cetuximab which does not require a wash-out), and all other immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) within 2 weeks, prior to the first dose of study treatment.
9. Chemotherapy within 4 weeks (except for bis-chlorethynitrosurea (BCNU), which must have been completed a minimum of 6 weeks) prior to starting therapy.
10. Major surgery within 4 weeks prior to the first dose of study treatment. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and patients should be recovered.
11. Use of other investigational drugs within 2 weeks or 5 half-lives (whichever is longer) prior to study treatment administration
12. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms); additional risk factors for torsades de pointes (TdP) (e.g., a history of heart failure, family history of Long QT Syndrome, or active hypokalemia or uncorrectable electrolyte abnormality); significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, congestive heart failure (New York Heart Association Class III or IV) related to primary cardiac disease, uncontrolled ischemic or severe valvular heart disease; or any of the following within 6 months prior to the first dose of study treatment: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack.
13. Requirement for chronic immunosuppressive medication including systemic corticosteroids above the physiologic dose (defined as 20 mg/day prednisone or the equivalent).
14. Any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.
15. Known alcohol or drug abuse.
16. Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
17. Inability to swallow pills
18. Patients unwilling or unable to comply with the protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NRAS Mutant Melanoma | WT Melanoma
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3
Not completed — Early Termination of Study | 0 | 3

BASELINE CHARACTERISTICS:
Population: The study was terminated before more participants could be enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | NRAS Mutant Melanoma | WT Melanoma | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 3 | 3
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 3 | 3
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: response rate, will be compared with the historically reported response rate for the single agent trametinib in NRAS and BRAF/NRAS WT melenoma
Time Frame: 48 Months
Population: Study was terminated prior to analysis.
Arm/Group | NRAS Mutant Melanoma | WT Melanoma
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Survival (OS)
Description: Survival data will be collectedvia telephone or clinic visits every 3 months (+10 days) from the date of last treatment, and median will be estimated using Kaplan-Meier approach
Time Frame: 48 Months
Population: Study was terminated prior to analysis.
Arm/Group | NRAS Mutant Melanoma | WT Melanoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Short duration of study prior to termination.
Arm/Group | WT Melanoma
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03580382/Prot_SAP_000.pdf